CLINICAL TRIAL: NCT01340612
Title: Stenting in the Treatment of Large, Wide-necked or Recurring Intracranial Aneurysms
Brief Title: Stenting in the Treatment of Aneurysm Trial
Acronym: STAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE10.111
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Intracranial Aneurysm
Keywords: large aneurysm; wide-necked aneurysm; recurring aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coiling (Active Comparator): endovascular coiling with any type of currently approved coil (first or second generation)
  Interventions: Device: endovascular coiling with any type of currently approved coil (first or second generation)
- coiling plus stenting (Active Comparator): endovascular stenting with or without coiling. The stent may be any of the currently approved stents for intracranial aneurysms.
  Interventions: Device: endovascular coiling with any type of currently approved coil (first or second generation); Device: endovascular stenting with or without coiling. The stent may be any of the currently approved stents for intracranial aneurysms.

INTERVENTIONS:
Device: endovascular coiling with any type of currently approved coil (first or second generation) — Standard procedure for endovascular coiling.Coils may be bare Platinum coils or any so-called second generation coils such as but not restricted to Hydrocoil or Cerecyte
Device: endovascular stenting with or without coiling. The stent may be any of the currently approved stents for intracranial aneurysms. — Standard procedure for stenting. Addition of coils to the stent is left to the judgment of the treating physician
  Arms: coiling plus stenting

SUMMARY:
The STAT trial aims at comparing coiling versus coiling plus stenting in patients with aneurysms prone to recurrence, that is large aneurysms or recurring aneurysms after previous coiling or wide-necked aneurysms. The primary hypothesis is that the use of stenting in addition to coiling decreases the recurrence rate from 33% to 20% at 12 months as compared to coiling alone.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting at least one aneurysm candidate for coiling, with large (≥10mm), wide-necked (>4mm), or recurrent lesions after coiling (but not stenting) and judged by the neurovascular team to require elective treatment provided that this single lesion, and no other aneurysm, will be treated during the endovascular session to be the object of the trial
* The anatomy of the lesion is such that endovascular treatment is judged possible with or without stenting
* The endovascular physician is a priori content to use either type of technique
* The patient has not previously been randomized into the trial
* Treatment is elective
* Patient is 18 or older
* Life expectancy is more than 2 years
* Patient has given fully informed consent and has signed consent form

Exclusion Criteria:

* Other aneurysms requiring treatment during the same session
* Patients with associated cerebral arteriovenous malformations
* Patients with recently ruptured aneurysms
* When parent vessel occlusion is the primary intent of the procedure
* Any absolute contraindication to endovascular treatment, angiography, or anesthesia such as severe allergies to contrast or medications, including ASA and Clopidogrel
* Patients with recurring, previously stented aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-08-25 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of target aneurysm | 12 months
  rate of angiographic recurrence

SECONDARY OUTCOMES:
Rate of Procedural complications defined as number of subjects with reported peri-procedural Adverse Events | 30 days
  Periprocedural Adverse Events is any type of complication or Adverse Event reported during or in the 30 days following the intervention
Rate of mortality and morbidity defined as the number of subjects with a disabling neurological events as measured by a modified Rankin Score greater than 2 during the follow-up period | 12 months
  A morbid event is defined as any Adverse Event of any severity being possibly or probably related to the disease or the treatment
Overall morbidity and mortality given by the modified Rankin Score | 12 months
  Overall morbidity and mortality is defined as a change in modified Rankin Score relative to baseline
Incidence of in-stent stenosis defined as the number of subjects with a reduction in the luminal diameter of greater than 50% | 12 months
  luminal diameter will be evaluated by an independent Core Lab

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame
Locations (5):
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame, Montreal, Quebec
- CHRU de Brest (Brest University Hospital), Brest, France

REFERENCES:
- [Derived] Naggara O, Darsaut T, Trystram D, Tselikas L, Raymond J. Unruptured intracranial aneurysms: why we must not perpetuate the impasse for another 25 years. Lancet Neurol. 2014 Jun;13(6):537-8. doi: 10.1016/S1474-4422(14)70091-2. No abstract available. PMID 24849854
- [Derived] Darsaut TE, Raymond J; STAT Collaborative Group. The design of the STenting in Aneurysm Treatments (STAT) trial. J Neurointerv Surg. 2012 May;4(3):178-81. doi: 10.1136/neurintsurg-2011-010065. Epub 2011 Jun 23. PMID 21990519